CLINICAL TRIAL: NCT03594578
Title: Effects of a Prospective Thinking Intervention on Delay Discounting in Patients With Hormone-Responsive Breast Cancer
Brief Title: Prospective Thinking in Hormone-Responsive Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey Stein, Research Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2574
Record Dates: First submitted 2018-06-25; First posted 2018-07-20 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Hormone Receptor Positive Malignant Neoplasm of Breast

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an episodic future thinking group or a control group (episodic recent thinking), stratified by menopausal status and baseline level of delay discounting.
Who Masked: Participant
Masking Description: Participants assigned to both groups will be masked to experimental hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Episodic future thinking (Experimental): Participants will complete a guided interview designed to elicit a number of personalized events that are likely to occur during various future time frames (e.g., 1 day, 1 week, 3 months, 1 year, etc.), as well as text cues designed to prompt episodic future thinking (e.g., "In 3 months, I will be at my daughter's wedding"). Text cues will be presented during subsequent behavioral tasks and participants will be asked to think vividly about these events.
  Interventions: Behavioral: Episodic future thinking
- Episodic recent thinking (control) (Sham Comparator): Participants will complete a guided interview designed to elicit a number of personalized events that occurred in the recent past (e.g., earlier today, yesterday), as well as text cues designed to prompt episodic thinking (e.g., "Earlier today, I was playing tennis with my wife."). Text cues will be presented during subsequent behavioral tasks and participants will be asked to think vividly about these events.
  Interventions: Behavioral: Episodic recent thinking

INTERVENTIONS:
Behavioral: Episodic future thinking — Prospective thinking intervention
  Arms: Episodic future thinking
Behavioral: Episodic recent thinking — Sham episodic thinking
  Arms: Episodic recent thinking (control)

SUMMARY:
One factor that limits the effectiveness of adjuvant hormone therapy for breast cancer is medication nonadherence. Adherence to long-term medication regimens requires valuation of temporally distant outcomes. Thus, interventions that improve valuation of the future, a phenomenon known as delay discounting, may improve medication adherence in breast cancer treatment and improve survival. This study will investigate the acute efficacy of a prospective thinking intervention (episodic future thinking) for reducing delay discounting and improving valuation of future health in breast cancer patients. Patients will engage in either episodic future thinking or a control condition during completion of delay discounting tasks in which they choose between immediate and delayed outcomes.

DETAILED DESCRIPTION:
Globally, breast cancer is the most common cause of cancer death among women. The most common pathological subtype is hormone receptor positive breast cancer, which accounts for approximately 70% of all diagnoses. Adherence to adjuvant hormone therapy (HT), including selective estrogen receptor modulators and aromatase inhibitors, in the treatment of hormone responsive breast cancer decreases risk of recurrence and increases overall survival among women. Unfortunately, up to half of patients discontinue HT prematurely or administer HT less frequently than prescribed, which increases risk of disease recurrence and associated mortality. Understanding the mechanisms underlying nonadherence will allow for development of targeted interventions to improve breast cancer survival.

A defining characteristic of adjuvant HT is that it provides no short-term benefits and, instead, prevents disease recurrence only after years of sustained adherence. In contrast, the benefits of discontinuing HT are relatively immediate (e.g., avoidance of adverse side effects, such as hot flashes or arthralgia). Thus, adherence to HT requires one's behavior to be guided by temporally distant outcomes, as bias toward immediate gratification narrows the temporal window over which future costs and benefits can motivate behavior. Therefore, treatment adherence may be understood through the behavioral economic process of delay discounting (i.e. devaluation of delayed outcomes), which provides a measure of how individuals value the future. Accumulating evidence shows that delay discounting is associated with a wide variety of maladaptive health behaviors, including failure to seek routine medical screening for cancer and other illnesses. However, no work has yet examined associations between delay discounting and adherence to cancer treatment, generally, or breast cancer treatment, specifically. This gap in knowledge represents a challenge to the understanding of risk factors for cancer-related morbidity and mortality and may limit the efficacy of breast cancer treatment.

Accordingly, the present study will investigate the acute efficacy of an episodic future thinking (EFT) intervention for reducing discounting and improving valuation of future health in breast cancer patients. EFT is a form of prospection that involves mental simulation of events that might occur in one's future. To some extent, EFT is an innate human ability that guides decision-making (e.g., simulating the experience of an upcoming job interview or social event); however, populations who discount the future rapidly show deficits in this ability, considering the future infrequently and demonstrating low-quality EFT content (e.g., fewer contextual and sensory details). Thus, EFT interventions are designed to remediate this deficit and reduce bias toward immediate gratification by guiding individuals to both generate high-quality EFT content and prompting them to engage in EFT frequently. Prior laboratory-based research by the investigative team and others has shown that EFT both reduces delay discounting and improves a wide range of maladaptive health behaviors and outcomes contributing to the development of cancer and survival following diagnosis and treatment, including tobacco use and dietary and weight control. The present study seeks to extend these findings by demonstrating that EFT improves laboratory-based measures of delay discounting and valuation of future health in breast cancer patients. Demonstrating EFT's acute efficacy in the laboratory would suggest that EFT may be adapted in future grant proposals as a targeted, remotely delivered intervention to improve HT adherence and subsequent breast cancer survival.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Female
* Must have a history of hormone responsive breast cancer treated with curative intent and have been recommended/prescribed adjuvant HT (tamoxifen, anastrozole, letrozole or exemestane) by their physician.

Exclusion Criteria:

* Recurrent breast cancer
* Adjuvant hormone therapy is no longer medically appropriate/advisable
* Incapable/ without capacity to provide personal consent
* Suffers from cognitive or physical impairments which interfere with medication self- administration and/or participation in episodic thinking
* Receiving HT for metastatic disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility will be based on self-reported gender.
Enrollment: 89 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Delay discounting (monetary) | 1 day
  Discount rate, k, for delayed monetary rewards
Delay discounting (cancer recurrence) | 1 day
  Discount rate, k, for delayed cancer recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S Stein, PhD, Principal Investigator — Virginia Tech Carilion School of Medicine and Research Institute
Locations (1):
- Virginia Tech Carilion Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaughn JE, Ammermann C, Lustberg MB, Bickel WK, Stein JS. Delay discounting and adjuvant endocrine therapy adherence in hormone receptor-positive breast cancer. Health Psychol. 2021 Jun;40(6):398-407. doi: 10.1037/hea0001077. PMID 34323542